CLINICAL TRIAL: NCT03747614
Title: Ocular Micro-vascular Research Base on Functional Slip Lamp Biomicroscopy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jin Yuan, Principal Investigator, Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 81670826
Record Dates: First submitted 2017-11-30; First posted 2018-11-20 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Dry Eye Syndromes; Inflammation; Microvessels
MeSH Terms: conditions — Dry Eye Syndromes; Inflammation | interventions — Fluorometholone; Tacrolimus

STUDY DESIGN:
Intervention Model Description: subjects from zhongshan ophthalmic center
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dry eye group (Experimental): The recruitment of subjects met the criteria of DEWS. Each subject received treatment based on increasing severity according to the expert consensus for the treatment of DE inflammation. For moderate levels of severity, topical anti-inflammatory agents (0.1% Fluorometholone) were administered twice daily and then gradually less frequently until inflammation was controlled. For severe DE, the approach was similar to that of the moderate level but with an increased concentration and treatment frequency of the anti-inflammatory agents (0.1% Fluorometholone, 4 times daily). Topical 0.05% tacrolimus twice daily when DE was extremely severe. Functional Slit-Lamp Biomicroscopy were administrated to collected data from this group.
  Interventions: Drug: Fluorometholone; Device: Functional Slit-Lamp Biomicroscopy
- Control group (Experimental): Normal health subject without drug intervention, Functional Slit-Lamp Biomicroscopy were administrated to collected data from this group.
  Interventions: Device: Functional Slit-Lamp Biomicroscopy

INTERVENTIONS:
Drug: Fluorometholone — Fluorometh010neEyeDrops:
  Brand names: Allergan Pharmaceuticals Ireland, Serial number: J20130061, NDC 60758-880-05. Tacrolimus Brand names: Senju Pharmaceutical Co., Ltd. Fukusaki Plant Serial number: H20130452
  Other Names: Tacrolimus
  Arms: Dry eye group
Device: Functional Slit-Lamp Biomicroscopy — A traditional slit lamp (HAAG-STREIT SWISS MADE 900.7.2.34925) was used, and a digital camera (Canon 60D. Canon Inc, Melville, NY) was attached via an inherent camera port. Custom software was used to measure the conjunctival microvascular BFV and vessel diameter using a protocol that has been previously described in detail. At baseline, video clips were recorded on six fields of the bulbar conjunctiva, which was approximately 1 mm from the limbus. During the follow-up visits, attention was given to relocating the vessel segments for these 6 fields.

SUMMARY:
Dry eye disease (DED), as one of the most common ocular surface diseases that affecting visual acuity, is highly associated with ocular surface inflammation. Until now, there is no accurate quantization index system to evaluate real-time ocular surface inflammation. Besides, an individualized therapy for ocular surface inflammation is also badly needed. As we all know, conjunctival congestion is one of the important clinical appearance of ocular surface inflammation. Hence, we suggest that several specific microvascular indexes could measure the change of ocular surface inflammation. Our program is aiming to investigate the correlation between inflammatory factors and blood flow velocity as well as microvascular distribution detecting from bulbar conjunctiva through our own devices and software.Futhermore, we tend to compare ocular surface microvascular indexes and microvascular distribution in normal people and dry eye patients in order to establish a database for Chinese people. By confirming the relationship between ocular surface microvascular indexes and ocular inflammation, we hope to set up new diagnostic criteria for ocular inflammation and an individualized therapeutic regimen based on ocular surface microvascular indexes. Finally, we want to establish a precision diagnostic and therapeutic pattern for dry eye disease.

DETAILED DESCRIPTION:
Dry eye (DE) is a growing public health concern that affects not only the visual function but also the quality of life of patients. In 2017, the International DE Study Workshop (DEWSII) adjusted the definition of DE by particularly emphasizing the inflammation in the ocular surface, and this adjustment represented a major shift in the understanding of dry eye disease (DED) pathogenesis and the facilitation of DED treatment.1,2 The recurrence of chronic and low-grade inflammation plays an important role in long-term disease progression and gradually deteriorates the ocular surface.3 Previous studies have concluded that the inflammatory response is involved in the pathological process of DE.4-7 The concentrations of IL-1α and mature IL-1ß in the tear fluid are increased.4,5 The activity of MMP-9, a suggested biomarker associated with ocular surface diseases including DE, is significantly elevated in Meibomian gland dysfunction (MGD), Sjögren's syndrome (SS) and aqueous tear deficiency (ATD).6 Other studies have indicated that inflammatory mediators such as IL-6, IL-8 and TNFα are expressed proportionally to the severity of DE symptoms, indicating the involvement of inflammation.7 The identification of inflammation as a major factor in DE informs the treatment strategy, including anti-inflammatory medication, which results in improvements to the ocular surface condition and to ocular comfort in DED patients.8,9 A series of studies have demonstrated improvements in the subjective and objective signs and symptoms of DE after anti-inflammatory and immunomodulatory therapies.8-11 To monitor the status of ocular surface inflammation and the ocular surface condition, traditional assessments, namely, evaluation of conjunctival hyperemia12 and corneal fluorescein staining using a slit lamp biomicroscope, are used. However, these methods are subjective and volatile and may not be sensitive indicators of the disease stage and treatment efficacy.13 A number of new tests have been used to distinguish inflammation.13-15 These new technologies include corneal confocal microscopy,15 conjunctival impression cytology16 and inflammatory tear-film cytokine tests in research and in the clinic.17 These newly implemented techniques have several limitations. Corneal confocal microscopy is a structure-based instrument with a narrow view of 400 × 400 µm2 that is limited to localization and cell counting. Conjunctival impression cytology16 and inflammatory tear-film cytokine tests19 are not routinely used, possibly due to the invasiveness, high cost and discomfort of these techniques.5,18 Therefore, the development of new methodologies to noninvasively and subjectively evaluate the inflammation status of the ocular surface is crucial.

The microvascular system of the bulbar conjunctiva can be easily accessed. The release of inflammatory cytokines on the ocular surface can cause vasodilation, which may result in alterations to the conjunctival microcirculation.19 Cheung et al. used a computer-assisted intravital microscope to evaluate vasculopathies of the conjunctival vessels and identified microvascular abnormalities in patients with diabetes20 and in patients who wore contact lens.21 Schulze et al. have also performed 'evaluations of the redness of the bulbar conjunctiva using fractal analysis and photometry.22 However, these studies did not directly measure the microcirculation. The microcirculation is an important aspect of the vascular system, may directly represent the hemodynamic response to ocular surface inflammation and may exhibit more sensitivity for monitoring vascular responses to anti-inflammatory treatment. Recently, Jiang et al. developed a functional slit-lamp biomicroscope that could be used to measure the conjunctival blood flow velocity (BFV) and vessel diameter.23 The goal of the present study was to characterize the microvasculature and microcirculation in the bulbar conjunctiva of DE patients in response to anti-inflammatory treatment.

ELIGIBILITY:
Inclusion Criteria:

* age ≧ 18 years
* Ocular Surface Disease Index (OSDI) ≧ 12.
* A 5-min Schirmer I test (ST) result showing less than 5 mm of moisture on the strip.
* A noninvasive average tear-film break-up time (NI-avBUT) less than 5 s.

Exclusion Criteria:

* Patients were excluded if they had an eye infection, injury, non-DE ocular inflammation, ocular surgery within the last 6 months, or any concurrent treatment that might interfere with the interpretation of the study results (systemic corticosteroids, immunosuppressive therapy, or hormonal replacement therapy). Patients were also excluded if they had an uncontrolled disease, had a significant illness or were pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — The participant eligibility is based on self-representation of gender identity.
Enrollment: 20 (Estimated)
Dates: Start 2017-06-30 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Conjunctival microvascular blood flow velocity | Baseline
  Acheived by a traditional slit lamp (HAAG-STREIT SWISS MADE 900.7.2.34925) with a digital camera (Canon 60D. Canon Inc, Melville, NY) and a custom software.
Conjunctival microvascular blood flow velocity | 30 days after commencement of treatment
  Acheived by a traditional slit lamp (HAAG-STREIT SWISS MADE 900.7.2.34925) with a digital camera (Canon 60D. Canon Inc, Melville, NY) and a custom software.
Conjunctival microvascular blood flow velocity | 60 days after commencement of treatment
  Acheived by a traditional slit lamp (HAAG-STREIT SWISS MADE 900.7.2.34925) with a digital camera (Canon 60D. Canon Inc, Melville, NY) and a custom software.
Conjunctival microvascular diameter | Baseline
  Acheived by a traditional slit lamp (HAAG-STREIT SWISS MADE 900.7.2.34925) with a digital camera (Canon 60D. Canon Inc, Melville, NY) and a custom software.
Conjunctival microvascular diameter | 30 days after commencement of treatment
  Acheived by a traditional slit lamp (HAAG-STREIT SWISS MADE 900.7.2.34925) with a digital camera (Canon 60D. Canon Inc, Melville, NY) and a custom software.
Conjunctival microvascular diameter | 60 days after commencement of treatment
  Acheived by a traditional slit lamp (HAAG-STREIT SWISS MADE 900.7.2.34925) with a digital camera (Canon 60D. Canon Inc, Melville, NY) and a custom software.
Conjunctival microvascular blood flow rate | Baseline
  Acheived by a traditional slit lamp (HAAG-STREIT SWISS MADE 900.7.2.34925) with a digital camera (Canon 60D. Canon Inc, Melville, NY) and a custom software.
Conjunctival microvascular blood flow rate | 30 days after commencement of treatment
  Acheived by a traditional slit lamp (HAAG-STREIT SWISS MADE 900.7.2.34925) with a digital camera (Canon 60D. Canon Inc, Melville, NY) and a custom software.
Conjunctival microvascular blood flow rate | 60 days after commencement of treatment
  Acheived by a traditional slit lamp (HAAG-STREIT SWISS MADE 900.7.2.34925) with a digital camera (Canon 60D. Canon Inc, Melville, NY) and a custom software.
The hyperemia index | Baseline
  The hyperemia index (HI) was measured by determining the percentage of conjunctival microvascular area in the conjunctiva automatically.26 The subjects were required to keep their eyes open and focus on the illuminated ring in front. Three consecutive readings were recorded, and the median was used. All data were recorded and analyzed with TF-scan software in the system.
The hyperemia index | 30 days after commencement of treatment
  The hyperemia index (HI) was measured by determining the percentage of conjunctival microvascular area in the conjunctiva automatically.26 The subjects were required to keep their eyes open and focus on the illuminated ring in front. Three consecutive readings were recorded, and the median was used. All data were recorded and analyzed with TF-scan software in the system.
The hyperemia index | 60 days after commencement of treatment
  The hyperemia index (HI) was measured by determining the percentage of conjunctival microvascular area in the conjunctiva automatically.26 The subjects were required to keep their eyes open and focus on the illuminated ring in front. Three consecutive readings were recorded, and the median was used. All data were recorded and analyzed with TF-scan software in the system.

SECONDARY OUTCOMES:
Non-invasived tear-film break-up time | Baseline
  The system measures the tear-film break-up time (NI-BUT) by monitoring the Placido projection on the cornea and includes the noninvasive first tear-film break-up time (NI-fBUT) and NI-avBUT. NI-fBUT and NI-avBUT were the measured times of the first and half-area breaks in the tear film between the full opening of the eyelids after 2 complete blinks.
Non-invasived tear-film break-up time | 30 days after commencement of treatment
  The system measures the tear-film break-up time (NI-BUT) by monitoring the Placido projection on the cornea and includes the noninvasive first tear-film break-up time (NI-fBUT) and NI-avBUT. NI-fBUT and NI-avBUT were the measured times of the first and half-area breaks in the tear film between the full opening of the eyelids after 2 complete blinks.
Non-invasived tear-film break-up time | 60 days after commencement of treatment
  The system measures the tear-film break-up time (NI-BUT) by monitoring the Placido projection on the cornea and includes the noninvasive first tear-film break-up time (NI-fBUT) and NI-avBUT. NI-fBUT and NI-avBUT were the measured times of the first and half-area breaks in the tear film between the full opening of the eyelids after 2 complete blinks.
Corneal Fluorescein Staining | Baseline
  Fluorescein was administered into the conjunctival sac under a cobalt blue light from the slit lamp. Corneal epithelial cell disruption was measured via corneal staining (National Eye Institute (NEI) scale, 5 areas of the cornea assessed (central, temporal, nasal, superior, and inferior), and the scores were assigned per a 0-8 scale for each area (total 40). Tear production was measured with Schirmer strips without anesthesia.
Corneal Fluorescein Staining | 30 days after commencement of treatment
  Fluorescein was administered into the conjunctival sac under a cobalt blue light from the slit lamp. Corneal epithelial cell disruption was measured via corneal staining (National Eye Institute (NEI) scale, 5 areas of the cornea assessed (central, temporal, nasal, superior, and inferior), and the scores were assigned per a 0-8 scale for each area (total 40). Tear production was measured with Schirmer strips without anesthesia.
Corneal Fluorescein Staining | 60 days after commencement of treatment
  Fluorescein was administered into the conjunctival sac under a cobalt blue light from the slit lamp. Corneal epithelial cell disruption was measured via corneal staining (National Eye Institute (NEI) scale, 5 areas of the cornea assessed (central, temporal, nasal, superior, and inferior), and the scores were assigned per a 0-8 scale for each area (total 40). Tear production was measured with Schirmer strips without anesthesia.
Schirmer I test | Baseline
  A meansurement of tear production with Schirmer strips and anaesthesia.
Schirmer I test | 30 days after commencement of treatment
  A meansurement of tear production with Schirmer strips and anaesthesia.
Schirmer I test | 60 days after commencement of treatment
  A meansurement of tear production with Schirmer strips and anaesthesia.

CONTACTS AND LOCATIONS:
Locations (1):
- Wan Chen, Guangzhou, Guangdong, China